

## RealGiDo

CTR display plan

RealGiDo: Real-world data on Gi(I)otrif® dose adjustment in first-line treatment, TKI-naïve, advanced non-small cell lung cancer patients with EGFR activating mutations

**Project No:** 5311000\_NIS RealGiDo

**Medication:** Gi(I)otrif <sup>®</sup>

**Dokument ID:** TechnicalSAP\_RealGiDo\_Final\_v1.1\_2018-01-17.docx

**Version:** Final 1.1

**Date:** 17.01.2018

Sponsor: Boehringer Ingelheim Pharma GmbH & Co. KG

Binger Straße 173

D-55216 Ingelheim am Rhein

**Author:** 

Protocol (Version, Date): Final version 1.0, 01.03.2016

## **Tables of contents**



The following tables, listings and figures are planned. The checked fields show the programmer where the parameter to be analysed may be found and will not appear in the report. In this context, the variable before the point displays the dataset and the variable after the point stands for the field name within the corresponding dataset. Take note, that the variable before the point must be always reported again as first term after the point, e.g. patient.birthyear stands for the field patient.patient\_birthyear in the eCRF.

Final 1.0, 29.11.2017 2 / 34

## 1 Methods for calculation of derived variables

<u>Age at registration:</u> Year of registration [patient.birthyear] – Year of birth [registration.registered\_at]

<u>Drug-related AE:</u> All AE with relationship to Gi(I)otrif<sup>®</sup> [ae.gilotref\_relation\_1='yes']

<u>Time on treatment:</u> Date of last administration [endofobservation.date] - Date of first administration of Gi(I)otrif<sup>®</sup> [baseline.date]. For patients still on treatment, time on treatment will be censored at the date of data collection.

<u>Time to progression (TTP):</u> First date of progression [min(endofobservation.radio\_date, endofobservation.clinic\_date)] - Date of first administration of Gi(I)otrif<sup>®</sup> [baseline.date]. Patients not known to have a progression will be censored with the date of last contact. For patients still on treatment and without progression, time to progression will be censored at the date of data collection. For patients who stopped treatment and without progression or progression date missing, time to progression will be censored on the last contact date.

## Missing / Incompete AE Onset Dates:

For each missing / incomplete AE onset date, an interval (INT\_START, INT\_END) is defined. The true unkniown analysis start date of the AE is assumed to be within this interval. If the AE onset date is completely missing INT START will be Min(AE end date, Date of informed consent) and INT END will be Min(AE end date, Date of last visit). If only the year of the AE onset date is non-missing INT\_START will be Min(AE end date, 01 JAN of the reported year) and INT END will be Min(AE end date, 31 DEC of the reported year). If only year and month of the AE onset date are non-missing INT START will be Min(AE end date, 01 of the reported month) and INT END will be Min(AE end date, Last date of the reported month). Completely missing AE end dae will not be considered in this derovation step. Partially missing AE end date (i.e., year and month are non-missing or only year is non-missing) will be temporarily assigned the largest possible date in the observed year or month and year in this derivation step. After this the imputed AE onset dates will be derived based on the intervals (INT START, INT END). If the date of first drug administration is within the interval [INT\_START, INT\_END] then the imputed AE onset date will be the date of drug administration. If the date of first drug administration is before INT START then the imputed AE onset date will equal INT\_START. If the date of first drug administration is after INT END or missing then the imputed AE onset date equals INT END.

Final 1.0, 29.11.2017 3 / 34

Final 1.0, 29.11.2017 4 / 34



Final 1.0, 29.11.2017 5 / 34



Final 1.0, 29.11.2017 6 / 34



Final 1.0, 29.11.2017 7 / 34



Final 1.0, 29.11.2017 8 / 34





















Final 1.0, 29.11.2017 18 / 34



Final 1.0, 29.11.2017 19 / 34



Final 1.0, 29.11.2017 20 / 34



Final 1.0, 29.11.2017 21 / 34



Final 1.0, 29.11.2017 22 / 34

23 / 34



Final 1.0, 29.11.2017 24 / 34



Final 1.0, 29.11.2017 25 / 34



Final 1.0, 29.11.2017 26 / 34



Final 1.0, 29.11.2017 27 / 34



Final 1.0, 29.11.2017 28 / 34



Final 1.0, 29.11.2017 29 / 34



Final 1.0, 29.11.2017 30 / 34



Final 1.0, 29.11.2017 31 / 34





Final 1.0, 29.11.2017 33 / 34



Final 1.0, 29.11.2017 34 / 34